CLINICAL TRIAL: NCT05298631
Title: Comparing the Effects of Neck Stabilization Exercises Verses Dynamic Exercises Among Patients Having Nonspecific Neck Pain With Forward Head Posture- A Randomized Clinical Trial
Brief Title: Comparing the Effects of Neck Stabilization Exercises Verses Dynamic Exercises Among Patients Having Nonspecific Neck Pain With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Asma Batool, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABatool
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Non-specific Neck Pain
Keywords: Neck Aches; Isotonic Contractions; Muscle Strength; Rehabilitation Exercises; Treatment
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: it is a randomized clinical trial. total 60 patients will be recruited 30 in each group. both groups are treatment group. treatment of group 1 is stabilization exercises and group 2 is dynamic exercises. patients are allocated randomly randomization is done by computer generated software sheet
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be blinded to the treatment provided to both treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1: stabilization exercises (Experimental): stabilization exercises
  1. Chin tuck
  2. Cervical extension
  3. Shoulder shrugs
  4. Shoulder rolls
  5. Scapular retraction (15 repetitions 1 set) with TENS(10 mins before each session for 10 min at the back of the neck), stretching of trapezius, Pectorals minor, sternocleidomastoid, levator scapulae (5 rep 10 sec hold 1 set in both sides ) and cold pack (10 min at the back of neck at the end of each session)
  Interventions: Other: Stabilization exercises
- Treatment group 2: dynamic exercises (Active Comparator): dynamic exercises
  1. Cervical extension-dynamic isometric.
  2. Cervical Flexion-Dynamic isometric.
  3. Chest flies exercises (15 repetitions 1 set) with TENS(10 mins before each session for 10 min at the back of the neck), stretching of trapezius, Pectorals minor, sternocleidomastoid, levator scapulae (5 rep 10 sec hold 1 set in both sides ) and cold pack (10 min at the back of neck at the end of each session)
  Interventions: Other: Dynamic exercises

INTERVENTIONS:
Other: Stabilization exercises — The activation of deep cervical muscle to reduce the activity of surface muscles is known as stabilization exercises
  Arms: Treatment group 1: stabilization exercises
Other: Dynamic exercises — The exercises in which muscle tension remains constant but muscle length changes is known as dynamic exercises
  Arms: Treatment group 2: dynamic exercises

SUMMARY:
the objective of this randomized clinical trial is to compare the effectiveness of neck stabilization exercises versus neck dynamic exercises in patients having non specific neck pain with forward head posture for pain intensity, correction of forward head posture, increasing Range of movement and decrease functional disability. the study is being conducted at physiotherapy department of institute of physical medicine and rehabilitation (Dow university of health sciences) total 60 patients with non specific neck pain with forward head posture recruited by non-probability sampling technique initially screening done by consultant physicians who is blinded to the treatment given to patients. patient are included in study who fulfill inclusion criteria and sign the consent form. patients then randomly allocated to both treatment groups using computer generated randomization sheet. baseline assessment is taken at first session after providing 9 treatment of stabilizing exercises to group1 and dynamic exercises to group 2 session post assessment will be done on goniometry, NDI, VAS and plumb line at last session at third week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonspecific neck pain more than 3 weeks less than 6 months.
* Patients with forward head posture on plumb line assessment.
* Pain on VAS moderate 4-7
* NDI score with moderate; 50-64%.
* Age ranges from 18-40.

Exclusion Criteria:

* Previous history of any accident (whiplash), fracture, tumor etc.
* Patients not willing to participate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity with Visual analog scale (VAS) in cm | Baseline and 3 weeks
  VAS will be used for assessment of pain intensity on 10 cm straight line with marking from 0 to 10 (0 means no pain and 10 means worst pain possible) patients pain is recorded at baseline at the start of 1st session than change in pain intensity (decrease) will be assessed at the end of 9th session at week 3.
Change in disability with Neck disability index questionnaire (NDI) scores | Baseline and 3 weeks
  NDI will be used for the assessment of disability due to neck pain. NDI is a ten item questionnaire each question has 6 responses from 0 no disability to 5 complete disability (score of less than 4 indicates no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, and scores greater than 35 complete disability) used to assess disability associated with neck pain and whiplash injury. patients disability is recorded at baseline at the start of 1st session than change in disability (decrease) will be assessed at the end of 9th session at week 3.
Change in neck range of motions with goniometer in degrees | Baseline and 3 weeks
  Goniometry will be used for the assessment of change in available range of motion of around neck joint in degrees. the therapist assess the range of motion using goniometer in flexion, extension, lateral flexion(right), lateral flexion(left), rotation(right), rotation(left). patients ROM is recorded at baseline at the start of 1st session than change in ROM (increase) will be assessed at the end of 9th session at week 3.
Change in ear position with reference to shoulder Plumb line measurement in inches | Baseline and 3 weeks
  Plumb line measurement will be used for the assessment of forward head posture using body landmarks such as ear lobe or mastoid process and shoulder alignment in inches. patients forward head is recorded at baseline at the start of 1st session than change in forward head (postural correction) will be assessed at the end of 9th session at week 3.

CONTACTS AND LOCATIONS:
Overall Officials: Aftab Ahmed Mirza Baig, MSAPT, Study Director — Sindh Institute of Physical Medicine and Rehabo; Rabail Rani Soomro, MSPT, Study Director — Sindh Institute of Physical Medicine and Rehabilitation
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batool A, Soomro RR, Baig AAM. Comparing the effects of neck stabilization exercises versus dynamic exercises among patients having nonspecific neck pain with forward head posture: a randomized clinical trial. BMC Musculoskelet Disord. 2024 Sep 4;25(1):707. doi: 10.1186/s12891-024-07749-8. PMID 39232708